CLINICAL TRIAL: NCT07011069
Title: Comparison of the Efficacy of Rhomboid Intercostal and Subserratus Plane Block (RISS) Versus Erector Spinae Plane (ESP) Blocks in Video-Assisted Thoracoscopic Surgery (VATS) for Postoperative Pain Management and Respiratory Function
Brief Title: Rhomboid Intercostal and Subserratus Plane Block vs Erector Spinae Plane Block in Video-Assisted Thoracoscopic Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bursa City Hospital (Other Government)
Responsible Party: Principal Investigator, Hande Gurbuz, Assoc. Prof., MD, PhD, Bursa City Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2024-11/4 24-AKD-209
Record Dates: First submitted 2025-05-23; First posted 2025-06-08 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-05

CONDITIONS: Video Assisted Thoracoscopic Surgery; Regional Block for Pain Control; Regional Blocks; Pulmonary Functions

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients who received ESP block (Active Comparator): Those who received the erector spinae plane block for postoperative pain management
  Interventions: Procedure: ESP block group
- Patients who received RISS block (Active Comparator): Those who received the rhomboid intercostal subserratus plane block for postoperative pain management
  Interventions: Procedure: RISS block group

INTERVENTIONS:
Procedure: ESP block group — ESP blocks are performed for patients undergoing VATS.
  Arms: Patients who received ESP block
Procedure: RISS block group — RISS blocks are performed for patients undergoing VATS.
  Arms: Patients who received RISS block

SUMMARY:
To compare the rhomboid intercostal subserratus plane block with the erector spinae plane block regarding their analgesic efficacy and effects on respiratory function for patients undergoing video-assisted thoracoscopic surgery.

DETAILED DESCRIPTION:
Video-assisted thoracoscopic surgery (VATS) can be very painful and may lead to complications such as prolonged stays in intensive care, thromboembolic complications due to lack of early mobilization, chronic acute pain, and delirium if adequate analgesia is not provided. Therefore, using thoracic epidural, paravertebral, or regional blocks as part of multimodal analgesia is recommended to provide effective pain relief.

This study aims to compare the effects of the erector spinae plane block (ESP) and rhomboid intercostal subserratus plane block (RISS) on postoperative analgesia and the improvement of respiratory parameters in patients undergoing VATS.

The primary objective is to evaluate total analgesic consumption in the first 24 hours postoperatively. Secondary objectives include assessing active and dynamic pain scores, triflow performance, complications, and the length of hospital stays.

ELIGIBILITY:
Inclusion Criteria:

* Patients who will undergo VATS
* Who agrees to participate
* American Society of Anesthesiologists (ASA) physical status I, II, and III
* Elective surgery
* Age between 18 and 80 years

Exclusion Criteria:

* Local anesthetic allergy
* Who disagrees to participate
* ASA physical status IV and V
* Emergency surgery
* Hemorrhagic disease
* Thoracic vertebrae deformity
* Thoracic vertebrae surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-11-15 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Opioid consumption | Postoperative first 24 hours.
  Total opioid consumption within the first 24 hours in the postoperative period.

SECONDARY OUTCOMES:
Dynamic pain score | Postoperative first 24 hours.
  Postoperative pain scores during coughing and deep breathing are measured on a 10 cm scale, where "0" indicates no pain and "10" indicates the worst pain ever.
Resting pain score | Postoperative first 24 hours.
  Postoperative pain scores during rest are measured on a 10 cm scale, where "0" indicates no pain and "10" indicates the worst pain ever.
Pulmonary functions | Postoperative first 24 hours.
  Pulmonary functions are assessed using Triflow performance. Postoperative Triflow numbers (whether 1, 2, or 3 balls can be raised) for the patients are recorded.
Complications | Through study completion, an average of 1 year
  Complications regarding regional blocks and surgery (such as hematoma, pulmonary complications) are recorded.
Hospital stay time | Perioperatively
  The length of hospital stay is recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences, Bursa City Hospital, Bursa, Nilufer, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The data sets used in this research may be made available upon reasonable request to the corresponding author.
Supporting Information: Study Protocol, SAP
Time Frame: 2026 to 2027
Access Criteria: The data sets used in this research may be made available upon reasonable request to the corresponding author.

REFERENCES:
- [Background] Forero M, Rajarathinam M, Adhikary S, Chin KJ. Erector spinae plane (ESP) block in the management of post thoracotomy pain syndrome: A case series. Scand J Pain. 2017 Oct;17:325-329. doi: 10.1016/j.sjpain.2017.08.013. Epub 2017 Sep 12. PMID 28919152
- [Background] Elsharkawy H, Maniker R, Bolash R, Kalasbail P, Drake RL, Elkassabany N. Rhomboid Intercostal and Subserratus Plane Block: A Cadaveric and Clinical Evaluation. Reg Anesth Pain Med. 2018 Oct;43(7):745-751. doi: 10.1097/AAP.0000000000000824. PMID 30169476
- [Background] Hsieh MJ, Wang KC, Liu HP, Gonzalez-Rivas D, Wu CY, Liu YH, Wu YC, Chao YK, Wu CF. Management of acute postoperative pain with continuous intercostal nerve block after single port video-assisted thoracoscopic anatomic resection. J Thorac Dis. 2016 Dec;8(12):3563-3571. doi: 10.21037/jtd.2016.12.30. PMID 28149550